CLINICAL TRIAL: NCT00393263
Title: A Double-Blind, Parallel-group Trial of Topical Pimecrolimus Cream 1% (Elidel®) Versus Clobetasol 0.05% Cream for the Treatment of Vulvar Lichen Sclerosus
Brief Title: Clobetasol Versus Pimecrolimus for Vulvar Lichen Sclerosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Center for Vulvovaginal Disorders (Other)
Collaborators: Novartis (Industry)
Responsible Party: Principal Investigator, Andrew T. Goldstein, MD, Director, Center for Vulvovaginal Disorders
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CASM981C US40
Record Dates: First submitted 2006-10-25; First posted 2006-10-27 (Estimated); Last update posted 2014-05-12 (Estimated); Status verified 2014-05

CONDITIONS: Lichen Sclerosus
MeSH Terms: conditions — Lichen Sclerosus et Atrophicus | interventions — pimecrolimus; Clobetasol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- 1 (Experimental): pimecrolimus
  Interventions: Drug: pimecrolimus and clobetasol
- 2 (Active Comparator): clobetasol
  Interventions: Drug: clobetasol 0.05% cream

INTERVENTIONS:
Drug: pimecrolimus and clobetasol
  Arms: 1
Drug: clobetasol 0.05% cream — twice daily for three months
  Arms: 2

SUMMARY:
Lichen sclerosus (LS) is a skin condition of the external genitals (vulva) of women. LS causes vulvar itching, pain, and burning. In addition, LS causes scarring of the vulva which may cause significant sexual dysfunction or pain. Lastly, 4-6% of women with LS will develop vulvar cancer.

The current "gold standard" treatment for lichen sclerosus is ultra-potent topical corticosteroids. When properly administered, topical ultra-potent corticosteroids help to resolve the symptoms of itching and burning and can prevent further vulvar scarring. In addition, proper treatment reverses the underlying inflammation of LS, and preliminary data shows that the risk of cancer also declines. While effective, topical corticosteroids have serious local and systemic side effects that include thinning of the skin, superimposed fungal infections, and suppression of the adrenal gland.

Elidel 1% cream is a new type of medication that has been approved by the FDA for the treatment of eczema. In theory, Elidel should also treat LS without the serious side effects that accompany corticosteroids. Therefore, this study is designed to compare the effectiveness and safety of a topical corticosteroid (clobetasol) versus Elidel 1% cream for the treatment of LS.

DETAILED DESCRIPTION:
Lichen sclerosus (LS) is a chronic cutaneous disorder affecting approximately one in seventy women. Presenting symptoms may include intense pruritis, pain, burning, and severe dyspareunia. The typical lesions of LS are white plaques and papules, often with areas of echymosis, excoriation, and ulceration. Often, LS causes destruction of the vulva architecture. In addition, 4-6% percent of women with LS will develop vulvar carcinoma. The histopathologic changes of LS are distinctive and make biopsy a very useful diagnostic tool. While there is no known cure for LS, the current gold standard treatment is ultra-potent corticosteroids. When properly administered, topical ultra-potent corticosteroids help to resolve the symptoms of pruritis and burning and can prevent further vulvar scarring. In addition, proper treatment reverses the underlying histopathologic changes of LS, and preliminary data shows that the risk of malignant transformation also declines. Although treatment with topical corticosteroids is effective, topical corticosteroids have serious local and systemic side effects, including dermal thinning, skin atrophy, superimposed fungal infections, rebound dermatitis, and adrenal insufficiency.

Pimecrolimus cream 1% (Elidel®, Novartis Pharmaceutical) is a topical calcineurin inhibitor that binds to macrophilin-12 and inhibits cytokine synthesis by T lymphocytes. Elidel has been approved by the FDA for the treatment of mild to moderate atopic dermatitis. In theory, as Elidel inhibits T lymphocytes, it should effectively treat lichen sclerosus. In addition, as Elidel does not inhibit keratinocytes, or affect collagen synthesis, it does not cause dermal atrophy. Therefore, Elidel may be an effective and safer alternative treatment for LS. This study is designed to compare the effectiveness and safety of Elidel 1% cream versus an ultra-potent corticosteroid (clobetasol 0.05% cream) for the treatment for vulvar LS.

ELIGIBILITY:
Inclusion Criteria:

* Female, 18 years or older.
* With a diagnosis of biopsy proven active vulvar lichen sclerosus.
* Signed written informed consent.
* Willingness and ability to comply with the study requirements.
* Negative urine pregnancy tests must be documented for all females of childbearing potential prior to enrollment.
* Two forms of birth control will be required for women with childbearing potential.
* IGA at baseline ≥1
* Subjects must have ≥ 4 or greater (on a 0 to 10 point scale) on at least one of the two visual analog scales (pruritus or pain/burning).

Exclusion Criteria:

* Who have received systemic immunosuppressants (e.g. corticosteroids) within 4 weeks prior to participation in the study.
* Who have been treated with topical therapy (e.g., topical corticosteroids, pimecrolimus, and tacrolimus) at the affected area within two weeks prior to participation in the study.
* Who are immunocompromised (e.g., lymphoma, AIDS, Wiskott-Aldrich Syndrome) or have an uncontrolled malignant disease.
* Who have a history of lymphoma
* Who have lympadenopathy
* Who have active vulvar herpes, molluscum, or condyloma
* Who suffer from systemic or generalized infections (bacterial, viral or fungal).
* Who have been diagnosed with lichen planus, psoriasis, candidiasis, intraepithelial neoplasia, or carcinoma of the vulva.
* Who have been diagnosed with diabetes mellitus or Netherton's syndrome.
* Menstruating females of childbearing potential who are not using two medically accepted methods of contraception during the study. Medically approved contraception may, at the discretion of the investigator, include abstinence.
* Women who are breastfeeding.
* Who had received an investigational drug within four weeks prior to the study or who intend to use other investigational drugs during the course of this study.
* Who are hypersensitive to pimecrolimus or clobetasol or any of the components of the creams.
* Patients with severe medical condition(s) that in the view of the investigator prohibits participation in the study.
* Who have a history of substance abuse or any factor, which limits the subject's ability to cooperate with the study procedures.
* Who are uncooperative, known to miss appointments (according to subjects' records) and are unlikely to follow medical instructions or are not willing to attend regularly scheduled visits.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2006-10; Primary Completion 2009-10 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
Change in inflammation | 3 months

SECONDARY OUTCOMES:
Pruritus | 3 months
Burning | 3 months
Pain | 3 months
Lichenification | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Andrew T Goldstein, MD, Principal Investigator — Center for Vulvovaginal Disorders
Locations (1):
- Center for VulvoVaginal Disorders, Washington D.C., District of Columbia, United States

REFERENCES:
- [Result] Goldstein AT, Marinoff SC, Christopher K. Pimecrolimus for the treatment of vulvar lichen sclerosus: a report of 4 cases. J Reprod Med. 2004 Oct;49(10):778-80. PMID 15568399
- [Result] Goldstein AT, Creasey A, Pfau R, Phillips D, Burrows LJ. A double-blind, randomized controlled trial of clobetasol versus pimecrolimus in patients with vulvar lichen sclerosus. J Am Acad Dermatol. 2011 Jun;64(6):e99-104. doi: 10.1016/j.jaad.2010.06.011. Epub 2011 Feb 25. PMID 21353334